CLINICAL TRIAL: NCT02319330
Title: Preventing & Treating HIV Comorbidities in India: Multi-tiered Strategy for Women
Acronym: MAHILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1301011297; R21MH100939 (NIH)
Record Dates: First submitted 2014-07-30; First posted 2014-12-18 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2019-08

CONDITIONS: HIV; Depression
Keywords: HIV; Adherence; Mental health; Depression; Women; Mobile phone technology; eHealth; India
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phone counseling intervention (Experimental): Treatment as usual (TAU) plus a nurse-delivered mobile phone counseling intervention delivered at weeks 1 to 12, 14, and 16 post-randomization.
  Interventions: Behavioral: Nurse-delivered mobile phone counseling intervention; Behavioral: Treatment as Usual
- Treatment as Usual (Active Comparator): Routine HIV clinic-based counseling
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Nurse-delivered mobile phone counseling intervention — Multi-dimensional, patient-centered counseling approach used to build patient-provider rapport, establish sources of support, and enable and empower problem solving to address inter-related, multi-tiered barriers to care.
  Arms: Phone counseling intervention
Behavioral: Treatment as Usual — Routine HIV clinic-based counseling

SUMMARY:
The overall objective of this project is to demonstrate that a low cost, cell phone-delivered intervention is a promising, feasible and acceptable way to improve the prevention and treatment outcomes of women in India who are affected by HIV and inter-related mental health and psychosocial risk factors.

DETAILED DESCRIPTION:
The overall objective of this project is to demonstrate that a low cost, cell phone-delivered intervention is a promising, feasible and acceptable way to improve the prevention and treatment outcomes of women in India who are affected by HIV and inter-related mental health and psychosocial risk factors. Over the past decade there have been dramatic improvements in HIV prevention and access to life-saving antiretroviral therapy (ART). Yet, deficits in adherence to the spectrum of HIV care pose significant barriers to success. Women are at a particular disadvantage. Gender inequality, physical and situational factors place many women at increased risk for HIV acquisition and poor mental health and interrelated psychosocial co-factors (depression, gender-discrimination, violence, lack of social support, etc.) that are well established correlates of poor adherence and retention in HIV care. Recent studies have shown alarmingly high rates of loss to follow-up for these women, particularly in the transition after delivery, between PMTCT and lifelong HIV care services. Preliminary work indicates that a theory-guided adherence phone intervention that can be easily integrated and sustained as a component of routine ART Centre services is well suited for the target population, but it needs to be adapted to the sociocultural context. Following initial formative work to refine the intervention for delivery in India, clinic nurses will be trained to deliver the intervention, and the feasibility, fidelity and preliminary efficacy of the novel application of the intervention will be evaluated in a randomized trial. After baseline assessment, women (n=120) will be randomly assigned to treatment as usual (TAU) or TAU plus the phone intervention (delivered over 16 weeks) and outcomes will be evaluated at 6, 14, 24, 36 weeks post-randomization. If the promising mobile phone intervention developed and pilot tested in this project shows promise in this Phase 1 study as we expect, the efficacy and cost of the intervention will then be evaluated in a large scale, multi-site study. If successful, an extremely practical approach will be available to improve the prevention and treatment outcomes of women with HIV and co-morbid mental health problems in India.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ women starting ART
* Willing to be contacted by mobile phone
* Speaks English or Hindi or Kannada
* Screens positive for depressive symptoms or psychosocial risk factors
* Able to provide informed consent

Exclusion Criteria:

* Unable to participate in study visits
* Any condition that, in the opinion of the site investigator, would compromise the candidate's ability to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Viral load | 6 months post-randomization
  HIV-1 RNA copies per millilitre of blood plasma

SECONDARY OUTCOMES:
Medication adherence | 6 weeks post-randomization
  Self-reported adherence to HIV medications
Mental health (Survey) | 6 weeks post-randomization
  Survey measures of symptoms of depression, anxiety and cognitive representation of illness
Medication adherence (Self-reported) | 14 weeks post-randomization
  Self-reported adherence to HIV medications
Medication adherence (Self-reported) | 24 weeks post-randomization
  Self-reported adherence to HIV medications
Medication adherence (Self-reported) | 36 weeks post-randomization
  Self-reported adherence to HIV medications
Mental health (survey) | 14 weeks post-randomization
  Survey measures of symptoms of depression, anxiety and cognitive representation of illness
Mental health | 24 weeks post-randomization
  Survey measures of symptoms of depression, anxiety and cognitive representation of illness
Mental health | 36 weeks post-randomization
  Survey measures of symptoms of depression, anxiety and cognitive representation of illness

OTHER OUTCOMES:
Feasibility and acceptability (Protocol specific tools) | 6 weeks post-randomization
  Protocol specific tools will be used to measure feasibility and user acceptability The assessment will include: 1) The ratio of eligible study participants to those enrolled; 2) Number of scheduled study visits completed at 6, 14, 24, and 36 weeks; 3) Attrition between baseline and follow-up; 4) Reason for premature drop-out; 5) Number of phone calls that were made on schedule; 6) Level of participation in intervention sessions including the total number sessions, number of sessions completed without break offs, number of break offs, length (minutes) of sessions; 7) Congruence of topic/content discussed on calls with protocol; 8) Patient and study nurse satisfaction with intervention content, mode of delivery, and protocol.
Feasibility and acceptability (Protocol specific tools) | 14 weeks post-randomization
  Protocol specific tools will be used to measure feasibility and user acceptability The assessment will include: 1) The ratio of eligible study participants to those enrolled; 2) Number of scheduled study visits completed at 6, 14, 24, and 36 weeks; 3) Attrition between baseline and follow-up; 4) Reason for premature drop-out; 5) Number of phone calls that were made on schedule; 6) Level of participation in intervention sessions including the total number sessions, number of sessions completed without break offs, number of break offs, length (minutes) of sessions; 7) Congruence of topic/content discussed on calls with protocol; 8) Patient and study nurse satisfaction with intervention content, mode of delivery, and protocol.
Feasibility and acceptability (Protocol specific tools) | 24 weeks post-randomization
  Protocol specific tools will be used to measure feasibility and user acceptability The assessment will include: 1) The ratio of eligible study participants to those enrolled; 2) Number of scheduled study visits completed at 6, 14, 24, and 36 weeks; 3) Attrition between baseline and follow-up; 4) Reason for premature drop-out; 5) Number of phone calls that were made on schedule; 6) Level of participation in intervention sessions including the total number sessions, number of sessions completed without break offs, number of break offs, length (minutes) of sessions; 7) Congruence of topic/content discussed on calls with protocol; 8) Patient and study nurse satisfaction with intervention content, mode of delivery, and protocol.
Feasibility and acceptability (Protocol specific tools) | 36 weeks post-randomization
  Protocol specific tools will be used to measure feasibility and user acceptability The assessment will include: 1) The ratio of eligible study participants to those enrolled; 2) Number of scheduled study visits completed at 6, 14, 24, and 36 weeks; 3) Attrition between baseline and follow-up; 4) Reason for premature drop-out; 5) Number of phone calls that were made on schedule; 6) Level of participation in intervention sessions including the total number sessions, number of sessions completed without break offs, number of break offs, length (minutes) of sessions; 7) Congruence of topic/content discussed on calls with protocol; 8) Patient and study nurse satisfaction with intervention content, mode of delivery, and protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Reynolds, PhD, Principal Investigator — Yale University; Prabha Chandra, MD, Principal Investigator — National Institute of Mental Health and Neuro Sciences (NIMHANS)
Locations (1):
- Belgaum ART Center, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds NR, Satyanarayana V, Duggal M, Varghese M, Liberti L, Singh P, Ranganathan M, Jeon S, Chandra PS. MAHILA: a protocol for evaluating a nurse-delivered mHealth intervention for women with HIV and psychosocial risk factors in India. BMC Health Serv Res. 2016 Aug 4;16(a):352. doi: 10.1186/s12913-016-1605-1. PMID 27491288
- [Derived] Satyanarayana VA, Duggal M, Jeon S, Singh P, Desai A, Chandra PS, Reynolds NR. Exploring the feasibility, acceptability and preliminary effects of a nurse delivered mhealth intervention for women living with HIV in South India: a pilot randomized controlled trial. Arch Womens Ment Health. 2024 Oct;27(5):751-763. doi: 10.1007/s00737-024-01462-0. Epub 2024 Apr 17. PMID 38630259
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730